CLINICAL TRIAL: NCT02436642
Title: AVERT Plus Post-Market Registry
Status: Terminated | Type: Observational
Why Stopped: business decision
Sponsor: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-6432
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AVERT Plus System

SUMMARY:
The devices used in this observational registry are the Osprey Medical Contrast Monitoring System (CMS) and the Osprey Medical AVERT Reflux Reduction System. Both products have CE Mark designations. The purpose of this registry is to evaluate the usability characteristics of the combined Osprey Medical AVERT System and the Contrast Monitoring System during normal clinical use.

DETAILED DESCRIPTION:
This is a prospective, single-center, non-randomized, single arm, observational registry of the AVERT System used in combination with the Contrast Monitoring System. Patients undergoing manual manifold injection coronary artery imaging for diagnostic or PCI procedures that utilize the AVERT System and the CMS will be included in this registry. Device use characteristics including, measurement of contrast media volume used, contrast media volume saved by the use of the AVERT System, evaluation of angiographic image quality, and physician feedback on device features and function will be obtained. All data will be collected on the day of the procedure and there will be no long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a coronary diagnostic or PCI procedure using manual manifold injection with the AVERT System and CMS according to the labeled indications for these devices.
* Patient consent to participate

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be included if they are scheduled for a coronary diagnostic or PCI procedure using manual manifold injection with the AVERT System and Contrast Monitoring System according to the labeled indications for these devices.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Contrast media volume usage | Day of procedure
  Compare cumulative contrast media volume usage as displayed by the CMS to volume estimation commonly performed in the catheterization laboratory

SECONDARY OUTCOMES:
Contrast media volume savings | Day of procedure
  Use the displayed volume savings function of the Contrast Monitoring System to determine the percent reduction in contrast media delivered to the patient due to the use of the AVERT System.
Angiographic image quality | Day of procedure
Physician feedback on device features | Day of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Desch, MD, Principal Investigator — Universitatsklinikum Schleswig-Holstein (Campus Lubeck)
Locations (1):
- Universitatsklinikum Schleswig-Holstein (Campus Lubeck), Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaye DM, Stub D, Mak V, Doan T, Duffy SJ. Reducing iodinated contrast volume by manipulating injection pressure during coronary angiography. Catheter Cardiovasc Interv. 2014 Apr 1;83(5):741-5. doi: 10.1002/ccd.25348. Epub 2014 Jan 7. PMID 24323791